CLINICAL TRIAL: NCT03360773
Title: Emotional Fluctuations in the Flow of Daily Life. Ecological Analysis of Depressive Symptoms in the General Population (FEDD).
Brief Title: Emotional Fluctuations in the Flow of Daily Life. Ecological Analysis of Depressive Symptoms in the General Population.
Acronym: FEDD
Status: Completed | Type: Observational
Sponsor: Universidad Autonoma de Madrid (Other)
Responsible Party: Principal Investigator, Marta Miret, Ph.D., Assistant Professor, Universidad Autonoma de Madrid
Other Study IDs: PI16/00177
Record Dates: First submitted 2017-11-07; First posted 2017-12-04 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Depression; Happiness; Personal Satisfaction
MeSH Terms: conditions — Depression; Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to analyze both depressive symptomatology and psychological well-being fluctuation in a day-to-day basis in the general population, in order to identify contextual determinants of the mood and well-being changes

DETAILED DESCRIPTION:
Introduction: The Experience Sampling Method is a research tool to study what people do and feel in their day to day. It allows to analyse temporal relationships between variables and has a high ecological validity.

Aim: To evaluate fluctuations of depressive symptoms and subjective well-being and to analyse the factors related to these fluctuations.

Methodology: Longitudinal study that will follow up for two weeks a representative sample of the population aged 18 to 65 years living in Madrid using the Experience Sampling Method. An interviewer will visit the participants at their home to carry out a structured interview on mental health and well-being and to install a mobile app on the smart phone of participants in order for them to fill out information about their emotional state during the following two weeks. Participants will use the smart phone screen to fill out a brief questionnaire about their feelings, the activities they are doing and the people with whom they are interacting. Multilevel analysis based on lineal hierarchical models will be employed for data analysis as well as methods based on machine learning.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Non-institutionalized resident in Madrid
* To own a smart phone

Exclusion Criteria:

* To present noticeable cognitive or other limitations that impede following the interview

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Residents of Madrid, Spain.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2018-03-10 (Actual); Primary Completion 2018-09-02 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Affect as measured by PANAS | 7 days
  Current experience of positive and negative emotions, along with the extent to which they are felt, by means of an adapted version of PANAS questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Miret García, Ph.D, Principal Investigator — Universidad Autonoma de Madrid
Locations (1):
- Universidad Autónoma de Madrid. Department of Psychiatry. School of Medicine, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided